CLINICAL TRIAL: NCT00874380
Title: Fiber Content of Hemodialysis Patients' Diet and it's Cardiovascular Implications.
Brief Title: Fiber Intake in an End Stage Renal Disease (ESRD) Population Followed Over 2 Years
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Suzanne El-Sayegh, Nephrology Attending, Assoc. Chair of Medicine, Northwell Health
Other Study IDs: 08-036
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Cardiovascular Outcome; Kalemia Control; Lipid Profile
Keywords: Fiber; Dialysis; Renal Replacement Therapy; Food Frequency Questionnaire; FFQ; Dietary counseling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: First describe the diet of a cohort of dialysis patients with focus on fiber content.
  Interventions: Other: Increasing total fiber intake in patient's diet

INTERVENTIONS:
Other: Increasing total fiber intake in patient's diet — Second counsel patients biweekly about their compliance with a high fiber diet, target being 25 to 30 gm of fiber a day.Follow them for a period of 2 years and assess if their is any significant decrease in their cardiovascular events and profile, in addition to assessing the effect of high fiber on kalemia.

SUMMARY:
Our research involves the detailed description of the content of the diet of x dialysis patients.

For our purpose we used a newly developed "food frequency questionnaire". This is the first validated questionnaire specific for dialysis patients and we were the first to use it.

Our special focus was the fiber content in the diet of our patient. Our thesis that they are way below the recommended guidelines for fiber intake was verified. Our follow will evaluate the effect of such at diet, mosTLy cardiovascular.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end stage renal disease on hemodialysis
* Patients who are able to give informed consent

Exclusion Criteria:

* Pregnant women.
* Cognitively impaired patients
* PEG feeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ESRD
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
cardiovascular event | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States